CLINICAL TRIAL: NCT05120518
Title: Post Mortem Tissue Donation of Pediatric Tumor Tissues and Cells
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Angela Waanders, Principle Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2019-2982
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue will be collected through a research tissue collection autopsy of the original tumor and other sites that are appropriate. Both tumor and normal cells will be collected during autopsy in addition to body fluids such cerebrospinal fluid (CSF), blood, bone marrow and skin biopsies for genomic testing.
  For brain tumor bio-specimens, through CBTN, we will store, analyze and share a large cohort of samples and within the repository protocol annotate and characterize using the latest genomic technologies. The information and materials collected will be used to support cross-disciplinary collaborations and coordinated research projects, focused on the molecular and cellular origins of children's tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients with cancer and non-cancer tumor types: Pediatric patients with cancer and non-cancer tumor types (solid, liquid, neuro-oncology and stem cell)
  Interventions: Other: Collection of post mortem tissue donation

INTERVENTIONS:
Other: Collection of post mortem tissue donation — Collection of post mortem tissue from pediatric participants with cancer and non-cancer tumor types from whom post mortem tissue donation and autopsy consent is obtained.

SUMMARY:
The objective of this study is to utilize all donated pediatric tumor tissues and cells obtained from autopsy to prospectively develop novel patient derived orthotopic xenograft (PDOX) mouse models as well as in vitro cell culture model systems for pediatric cancers, and also provide tissue samples to other researchers and organizations (eg, CBTN, DIPG Registry, COG).

DETAILED DESCRIPTION:
The objective of this study is to utilize all donated pediatric tumor tissues and cells obtained from autopsy to prospectively develop novel patient derived orthotopic xenograft (PDOX) mouse models as well as in vitro cell culture model systems for pediatric cancers, and also provide tissue samples to other researchers and organizations (eg, CBTN, DIPG Registry, COG).

This model system will then be subjected to 1) comprehensive histopathological and molecular characterizations during serial in vivo sub-transplantations; 2) cryopreserved for long term preservation of tumorigenicity; and 3) used for future biological studies and preclinical drug testing.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with cancer and non-cancer tumor types (solid, liquid, neuro-oncology)
* Signed consent for post mortem tissue donation and autopsy

Exclusion Criteria:

* Signed consent for post mortem tissue donation and autopsy not obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients with cancer and non-cancer tumor types (solid, liquid, neuro-oncology)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2029-08-14 (Estimated); Study Completion 2029-08-14 (Estimated)

PRIMARY OUTCOMES:
Procurement of pediatric cancer and non-cancer tumor tissue during autopsy with signed consent | Up to 5 years from procurement
  Procurement of pediatric cancer and non-cancer tumor tissue during autopsy with signed consent. Tissue will be collected through a research tissue collection autopsy of the original tumor and other sites that are appropriate. Samples of both tumor and normal cells will be collected in addition to body fluids such as cerebrospinal fluid (CSF), blood, bone marrow, and skin biopsies for genomic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Waanders, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
To provide samples and PHI to CBTN. Samples and data will be de-identified prior to placement in the CBTN Biorepository.
Supporting Information: Study Protocol, ICF
Time Frame: Starting August 2019
Access Criteria: The IPD for this study will be stored in the CBTN Biorepository. Samples and data will be de-identified prior to placement in the CBTN Biorepository. Researchers who have been granted access to the CBTN Biorepository will have access to the IPD for this study.

REFERENCES:
- [Background] Baker JN, Windham JA, Hinds PS, Gattuso JS, Mandrell B, Gajjar P, West NK, Hammarback T, Broniscer A. Bereaved parents' intentions and suggestions about research autopsies in children with lethal brain tumors. J Pediatr. 2013 Aug;163(2):581-6. doi: 10.1016/j.jpeds.2013.01.015. Epub 2013 Feb 19. PMID 23433673
- [Background] Broniscer A, Baker JN, Baker SJ, Chi SN, Geyer JR, Morris EB, Gajjar A. Prospective collection of tissue samples at autopsy in children with diffuse intrinsic pontine glioma. Cancer. 2010 Oct 1;116(19):4632-7. doi: 10.1002/cncr.25405. PMID 20589749
- [Background] Wiener L, Sweeney C, Baird K, Merchant MS, Warren KE, Corner GW, Roberts KE, Lichtenthal WG. What do parents want to know when considering autopsy for their child with cancer? J Pediatr Hematol Oncol. 2014 Aug;36(6):464-70. doi: 10.1097/MPH.0000000000000078. PMID 24309611
- [Background] Alabran JL, Hooper JE, Hill M, Smith SE, Spady KK, Davis LE, Peterson LS, Malempati S, Ryan CW, Acosta R, Spunt SL, Keller C. Overcoming autopsy barriers in pediatric cancer research. Pediatr Blood Cancer. 2013 Feb;60(2):204-9. doi: 10.1002/pbc.24320. Epub 2012 Sep 26. PMID 23015377
- [Background] Meeting Minutes: Enhancing Biobanking for Childhood Cancers, NCI, May 13, 2019
- See also: Related Info — http://www.cancer.gov
- See also: Related Info — http://genome.gov